CLINICAL TRIAL: NCT02979522
Title: An Open-Label Study of Brentuximab Vedotin + Adriamycin, Vinblastine, and Dacarbazine in Pediatric Patients With Advanced Stage Newly Diagnosed Hodgkin Lymphoma
Brief Title: A Study of Brentuximab Vedotin + Adriamycin, Vinblastine, and Dacarbazine in Pediatric Participants With Advanced Stage Newly Diagnosed Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C25004; 2015-004112-38 (EudraCT Number); U1111-1171-0984 (Registry Identifier: WHO); 2023-506415-18-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2016-11-11; First posted 2016-12-01 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hodgkin Disease
Keywords: Drug therapy, pediatric Hodgkin disease, frontline Hodgkin disease, advanced stage Hodgkin disease, pediatric lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD (Experimental): Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles.
  Interventions: Drug: Brentuximab vedotin; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine
- Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD (Experimental): Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles.
  Interventions: Drug: Brentuximab vedotin; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin infusion
  Other Names: Adcetris
Drug: Doxorubicin — Doxorubicin infusion
  Other Names: Adriamycin
Drug: Vinblastine — Vinblastine infusion
Drug: Dacarbazine — Dacarbazine infusion

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and anti-tumor activity, as well as confirm the recommended dose of brentuximab vedotin (ADCETRIS) in combination with a multiagent chemotherapy regimen, doxorubicin (Adriamycin), vinblastine, and dacarbazine, in pediatric participants with advanced stage newly diagnosed classical CD30+ Hodgkin Lymphoma (HL).

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin. Brentuximab vedotin is being tested to treat pediatric participants who have advanced stage, newly diagnosed, classical CD30+ HL. This study will assess the safety, tolerability, and anti-tumor activity, as well as recommended dose of brentuximab vedotin in combination with a multiagent chemotherapy regimen that is based on a current standard of care (SOC) first-line treatment regimen for newly diagnosed HL.

The study will enroll approximately 55 evaluable participants. The study will be conducted in 2 phases, Phase 1 and Phase 2. Phase 1 study will enroll at least 6 participants to determine the recommended dose. Once the recommended dose is identified additional participants will be enrolled into phase 2 so that the total number of evaluable participants will be at least 55, including participants treated at recommended dose in Phase 1. Participants will be enrolled to the following initial dose cohort with an option to explore a reduced dose cohort at 36 mg/m^2 if needed:

• Brentuximab vedotin 48 mg/m^2 in combination with doxorubicin, vinblastine, and dacarbazine.

This multi-center trial will be conducted in the United States, Italy, Brazil and Japan. The overall time to participate in this study is approximately 55 months, including the follow-up period. Participants will be followed for a maximum of 30 days following the last dose of protocol therapy for a follow-up assessment and will be followed for survival and disease status every 12 weeks for 12 months, and then every 24 weeks until death or study closure or for up to 2 years from the date of the last participant enrolled.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all the following inclusion criteria to be enrolled in the study:

1. Histologically confirmed CD30+ classical HL.
2. Advanced stage, newly diagnosed HL (Stage III and Stage IV disease).
3. Treatment-naive HL.
4. Have performance scores of greater than or equal to (>=) 50 for Lansky Play-performance or Karnofsky Performance Status.
5. Have bidimensional measurable disease as documented by radiographic technique per International Working Group (IWG) criteria.
6. Have adequate blood counts, renal and liver function as defined in the protocol.

Exclusion Criteria:

1. Nodular lymphocyte predominant HL.
2. Known active cerebral/meningeal disease, including signs or symptoms of progressive multifocal leukoencephalopathy (PML) or any history of PML.
3. Any sensory or motor peripheral neuropathy.
4. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications.
5. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks before the first study protocol therapy.
6. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin or any component of AVD.
7. Known human immunodeficiency virus positive.
8. Known hepatitis B surface antigen positive or known or suspected active hepatitis C infection, as determined by hepatitis B DNA or hepatitis C RNA, respectively, in blood.
9. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
10. Use of any strong or listed moderate cytochrome P450 (CYP) 3A4 inhibitors less than (<) 2 weeks before the first dose of protocol therapy (please refer to the Study Manual for an example list of prohibited CYP3A4 inhibitors).
11. Any of the following cardiovascular conditions or values within 6 months before the first dose of protocol therapy:

    * Shortening fraction of <27 percent (%) by echocardiogram or, if echocardiogram not feasible, ejection fraction of <50% by radionuclide angiogram (RNA or MUGA [multiple-gated acquisition scan]).
    * New York Heart Association Class III or IV heart failure.
    * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2029-09-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Brazil (6):
  - Hospital Sao Rafael S/A, Salvador, Estado de Bahia
  - Jardim das Americas, Paranã
  - INCA - Instituto Nacional de Cancer, Rio de Janeiro
  - GRAACC - Grupo de Apoio ao Adolescente e a Crianca com Cancer, São Paulo
  - ICr - Instituto da Crianca - HCFMUSP, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Italy (4):
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Pediatrico Bambino Gesu,UOC Onco-ematologia, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (2):
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Suri A, Mould DR, Song G, Kinley J, Venkatakrishnan K. Population Pharmacokinetics of Brentuximab Vedotin in Adult and Pediatric Patients With Relapsed/Refractory Hematologic Malignancies: Model-Informed Hypothesis Generation for Pediatric Dosing Regimens. J Clin Pharmacol. 2020 Dec;60(12):1585-1597. doi: 10.1002/jcph.1682. Epub 2020 Jun 28. PMID 32596842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced stage newly diagnosed, classical CD30+ Hodgkin Lymphoma (HL) took part in the study at 14 investigative sites in the United States, Italy, Brazil and Japan from 06 September 2017 to data cut-off date: 24 September 2021. This study is ongoing for Post-Treatment Follow-Up (which includes Progression-Free Survival Follow-Up [PFSFU] and Overall Survival Follow-Up [OSFU]) and optional Long-Term Safety Follow-up.
Pre-assignment Details: Participants with advanced stage newly diagnosed, classical CD30+ HL received brentuximab vedotin 48 mg/m^2 in combination with doxorubicin, vinblastine, and dacarbazine(A+AVD). Data for Phase 2 endpoints is reported for participants enrolled in Phase 2 only and for all treated in Phase 2, including Phase 1 participants.
Period: Overall Study
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Started | 8 | 51
Completed | 0 | 0
Not Completed | 8 | 51
Not completed — Post-Treatment Follow-up (PFSFU and OSFU) | 0 | 28
Not completed — Particpants Ongoing in Long-Term Safety Follow-Up | 8 | 23

BASELINE CHARACTERISTICS:
Population: The safety population included participants who had received at least 1 dose of any study drug (A+AVD regimen).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Total
Number analyzed (Participants) | 8 | 51 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (3.81) | 13.9 (2.88) | 13.7 (3.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 24 | 28
  Male | 4 | 27 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 21 | 23
  Not Hispanic or Latino | 6 | 26 | 32
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 3 | 3
  Black or African American | 0 | 12 | 12
  White | 8 | 26 | 34
  "Brown" or "Mulatto" | 0 | 9 | 9
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 10 | 12
  Japan | 0 | 2 | 2
  Italy | 5 | 10 | 15
  Brazil | 1 | 29 | 30
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 45.91 (18.867) | 49.91 (15.649) | 49.37 (16.000)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Recommended Dose of Brentuximab Vedotin in Combination With Doxorubicin, Vinblastine, and Dacarbazine in a Pediatric Population
Description: The recommended dose was determined after considering all safety data in phase 1 and assessing for dose limiting toxicities (DLTs) which are defined as the dose range at which less than or equal to (<=) 1 of 6 evaluable participants experience DLT within the defined observation period (Cycle 1 + 28 days). This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: From the first dose (Cycle 1) up to Day 56 (Cycle length=28 days)
Population: The DLT-evaluable population included participants who had received at least 1 dose of study drug therapy and experienced a DLT or no DLT during the DLT observation period. Participants who received granulocyte colony stimulating factor (G-CSF) during the DLT observation period were excluded from the DLT-Evaluable Population.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD: Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 56 days.
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 6
mg/m^2 | 48

2. Primary Outcome: Phase 1: Percentage of Participants Who Experienced Adverse Events (AEs) From the First Dose of Protocol Therapy Through 30 Days After Administration of the Last Dose of Protocol Therapy
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: From first dose in Cycle 1 Day 1 until 30 days after the last dose of study drug in Cycle 6 Day 15 (up to Cycle 7 Day 15) (Cycle length=28 days)
Population: The safety population included participants who had received at least 1 dose of any study drug (A+AVD regimen).
Measure: Number; unit: percentage of participants
Groups:
- Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD: Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles. Participants who received at least one dose of study in Phase 1 and continued to receive the study drug in Phase 2 were included in this arm group.
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 100

3. Primary Outcome: Phase 1: Percentage of Participants Who Experienced Serious Adverse Events (SAEs) From the First Dose of Protocol Therapy Through 30 Days After Administration of the Last Dose of Protocol Therapy
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. SAE is defined as any untoward medical occurrence that at any dose results in death, Is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, Is a congenital anomaly/birth defect, Is a medically important event.
Time Frame: as for outcome 2
Population: The safety population included participants who had received at least 1 dose of any study drug (A+AVD regimen).
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 13

4. Primary Outcome: Phase 2: Percentage of Participants Who Achieved a Complete Remission (CR) Per Independent Review Facility (IRF) Assessment Per International Working Group (IWG) Criteria at End of Treatment (EOT) Visit
Description: CR was defined as the disappearance of all evidence of disease as assessed by IRF as per IWG Criteria. The confidence interval was based on exact binomial distribution (Clopper-Pearson method). This outcome measure was planned to be assessed for all participants treated at the recommended dose in Phase 2. As prespecified in the statistical analysis plan (SAP) , data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: At end of treatment (EOT) visit 30 days after the last dose of study drug (at Month 7)
Population: Response-evaluable population included participants who received at least one dose of study drug, have measurable disease at baseline, and have at least one post-baseline disease assessment based on an independent review facility.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD: Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles. Participants enrolled in Phase 2 were included.
- Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD: Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles.
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 75 [60 to 86] | 76 [63 to 86]

5. Primary Outcome: Phase 2: Percentage of Participants Whose Disease Was Positron Emission Tomography (PET) Negative After 2 Cycles of Protocol Therapy Per IRF Assessment
Description: The Deauville score according to IRF assessment of response was used to evaluate the results of PET scans. PET negative after Cycle 2 was defined as an IRF Deauville score of (1 or 2 or 3). This outcome measure was planned to be assessed for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: From first dose of study drug up to Cycle 2 Day 25 (Each Cycle length=28 days)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 90 | 90

6. Primary Outcome: Phase 2: Percentage of Participants Who Achieved a Partial Remission (PR) Per IRF Assessment Per IWG Criteria at EOT Visit
Description: PR was defined as regression of measurable disease and no new sites as assessed by IRF as per IWG criteria. Percentage of participants in the response-evaluable population who achieved a partial response based on the IRF assessment at the EOT visit based on the IWG criteria are reported. The confidence interval was based on exact binomial distribution (Clopper-Pearson method). This outcome measure was planned to be assessed for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: At EOT visit 30 days after the last dose of study drug (at Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 12 [6 to 20] | 12 [5 to 23]

7. Primary Outcome: Phase 2: Percentage of Participants Who Achieved an Overall Response Rate (ORR) Per IRF Assessment Per IWG Criteria at EOT Visit
Description: Overall response rate was defined as the percentage of participants with CR or PR as assessed by IRF using IWG criteria. CR was defined as the disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new diseases. The confidence interval was based on exact binomial distribution (Clopper-Pearson method). This outcome measure was planned to be assessed for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: At EOT visit 30 days after the last dose of study drug (at Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 86 [74 to 94] | 88 [77 to 95]

8. Primary Outcome: Phase 2: Percentage of Participants Who Were Able to Complete 6 Cycles of Protocol Therapy at the Recommended Dose
Description: This outcome measure was planned to be assessed for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: From first dose of study drug up to Cycle 6 (Each Cycle length=28 days)
Population: The safety population included participants who had received at least 1 dose of any study drug (A+AVD regimen).
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 100 | 100

9. Secondary Outcome: Phase 1: Mean Maximum Observed Serum Concentration (Cmax) of Brentuximab Vedotin Total Conjugated and Therapeutic Antibody (TAb)
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: The PK population included participants with sufficient data to enable calculation of at least 1 PK parameter. Number analyzed is number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: microgram per milliliter(mcg/mL)
Groups:
- Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD: Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles.
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
microgram per milliliter(mcg/mL)
  Conjugate Brentuximab Vedotin at Cycle 1 Day 1 | 22.6 (1.51)
  Conjugate Brentuximab Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 6
  Conjugate Brentuximab Vedotin at Cycle 1 Day 15 | 23.1 (3.85)
  Conjugate Brentuximab Vedotin at Cycle 3 Day 1 | 26.7 (3.65)
  Conjugate Brentuximab Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 7
  Conjugate Brentuximab Vedotin at Cycle 3 Day 15 | 27.3 (7.14)
  TAb at Cycle 1 Day 1: number analyzed (Participants) | 7
  TAb at Cycle 1 Day 1 | 24.9 (3.84)
  TAb at Cycle 1 Day 15: number analyzed (Participants) | 6
  TAb at Cycle 1 Day 15 | 25.5 (5.28)
  TAb at Cycle 3 Day 1: number analyzed (Participants) | 6
  TAb at Cycle 3 Day 1 | 29.6 (4.05)
  TAb at Cycle 3 Day 15: number analyzed (Participants) | 6
  TAb at Cycle 3 Day 15 | 28.1 (7.45)

10. Secondary Outcome: Phase 1: Mean Maximum Observed Plasma Concentration (Cmax) of Monomethyl Auristatin E (MMAE)
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
nanogram per milliliter (ng/ml)
  Cycle 1 Day 1 | 5.51 (3.91)
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 2.08 (0.677)
  Cycle 3 Day 1 | 1.38 (0.514)
  Cycle 3 Day 15: number analyzed (Participants) | 7
  Cycle 3 Day 15 | 1.19 (0.366)

11. Secondary Outcome: Phase 1: Mean Area Under the Serum Concentration-Time Curve From Day 0 to Day 15 (AUC0-15) of Brentuximab Vedotin and TAb
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: The PK population included participants with sufficient data to enable calculation of at least 1 PK parameter, with data available for analyses. Number analyzed is number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: day*microgram per milliliter(day*mcg/mL)
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 7
day*microgram per milliliter(day*mcg/mL)
  AUC0-15d of Brentuximab Vedotin at Cycle 1 Day 1 | 42.3 (3.10)
  AUC0-15d of Brentuximab Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 6
  AUC0-15d of Brentuximab Vedotin at Cycle 1 Day 15 | 48.8 (5.83)
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 1 | 72.7 (27.8)
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 6
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 15 | 64.8 (13.5)
  AUC0-15d of TAb at Cycle 1 Day 1 | 80.6 (13.0)
  AUC0-15d of TAb at Cycle 1 Day 15: number analyzed (Participants) | 6
  AUC0-15d of TAb at Cycle 1 Day 15 | 103 (14.6)
  AUC0-15d of TAb at Cycle 3 Day 1: number analyzed (Participants) | 6
  AUC0-15d of TAb at Cycle 3 Day 1 | 127 (10.2)
  AUC0-15d of TAb at Cycle 3 Day 15: number analyzed (Participants) | 6
  AUC0-15d of TAb at Cycle 3 Day 15 | 128 (34.4)

12. Secondary Outcome: Phase 1: Mean Area Under the Plasma Concentration-Time Curve From Day 0 to Day 15 (AUC0-15) of MMAE
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day* nanogram per milliliter (day*ng/mL)
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 7
day* nanogram per milliliter (day*ng/mL)
  Cycle 1 Day 1 | 29.8 (21.2)
  Cycle 1 Day 15: number analyzed (Participants) | 3
  Cycle 1 Day 15 | 13.1 (2.99)
  Cycle 3 Day 1 | 8.88 (2.53)
  Cycle 3 Day 15: number analyzed (Participants) | 4
  Cycle 3 Day 15 | 7.17 (2.17)

13. Secondary Outcome: Phase 1: Median Time to Reach Cmax (Tmax) of Brentuximab Vedotin and TAb in Serum
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Cycle 1-6: Days 1 and 15 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: The PK population included participants with sufficient data to enable calculation of at least 1 PK parameter, with data available for analyses.
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
hour
  Tmax of Brentuximab Vedotin at Cycle 1 Day 1 | 1.00 [0.570 to 1.05]
  Tmax of Brentuximab Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 6
  Tmax of Brentuximab Vedotin at Cycle 1 Day 15 | 0.915 [0.580 to 1.00]
  Tmax of Brentuximab Vedotin at Cycle 3 Day 1 | 1.00 [0.630 to 1.17]
  Tmax of Brentuximab Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 7
  Tmax of Brentuximab Vedotin at Cycle 3 Day 15 | 0.830 [0.580 to 1.00]
  Tmax of TAb at Cycle 1 Day 1: number analyzed (Participants) | 7
  Tmax of TAb at Cycle 1 Day 1 | 1.00 [0.570 to 1.05]
  Tmax of TAb at Cycle 1 Day 15: number analyzed (Participants) | 6
  Tmax of TAb at Cycle 1 Day 15 | 0.915 [0.580 to 1.00]

14. Secondary Outcome: Phase 1: Median Time to Reach Cmax (Tmax) of MMAE in Plasma
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
hour
  Cycle 1 Day 1 | 44.9 [21.1 to 69.1]
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 43.1 [41.2 to 45.9]
  Cycle 3 Day 1 | 48.0 [42.3 to 66.9]
  Cycle 3 Day 15: number analyzed (Participants) | 7
  Cycle 3 Day 15 | 48.2 [20.8 to 67.0]

15. Secondary Outcome: Phase 1: Percentage of Participants Who Achieved a CR Per IRF Assessment Per IWG Criteria at EOT Visit
Description: CR was defined as the disappearance of all evidence of disease as assessed by IRF as per IWG Criteria. The confidence interval was based on exact binomial distribution (Clopper-Pearson method). This outcome measure was planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: At EOT visit 30 days after the last dose of study drug (at Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 88 [47 to 100]

16. Secondary Outcome: Phase 1: Percentage of Participants Who Achieved a PR Per IRF Assessment Per IWG Criteria at EOT Visit
Description: PR was defined as regression of measurable disease and no new diseases as per IWG Criteria based on IRF. The confidence interval was based on exact binomial distribution (Clopper-Pearson method). This outcome measure was planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: At EOT visit 30 days after the last dose of study drug (at Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 13 [1 to 53]

17. Secondary Outcome: Phase 1: Percentage of Participants Who Achieved an ORR Per IRF Assessment Per IWG Criteria at EOT Visit
Description: Overall response rate was defined as the percentage of participants with CR or PR as assessed by an IRF using IWG Revised Response Criteria. CR was defined as the disappearance of all evidence of disease and PR was defined as regression of measurable disease and no new sites. The confidence interval was based on exact binomial distribution (Clopper-Pearson method). This outcome measure was planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: At EOT visit 30 days after the last dose of study drug (at Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 100 [63 to 100]

18. Secondary Outcome: Phase 1: Percentage of Participants Whose Disease Was PET Negative After 2 Cycles of Protocol Therapy Per IRF Assessment
Description: The Deauville score according to IRF assessment of response was used to evaluate the results of PET scans. PET negative after Cycle 2 was defined as an IRF Deauville score of (1 or 2 or 3). This outcome measure was planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: From first dose of study drug up to Cycle 2 (Each Cycle length=28 days)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 88 [47 to 100]

19. Secondary Outcome: Phase 1: Percentage of Participants Whose Disease Was PET Positive After 6 Cycles of Protocol Therapy Per IRF Assessment
Description: The Deauville score according to IRF assessment of response was used to evaluate the results of PET scans. PET positive after Cycle 6 defined as an IRF Deauville score of (4 or 5). This outcome measure was planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: From first dose of study drug up to Cycle 6 (Each Cycle length=28 days)
Population: This outcome measure was planned to be assessed only for participants treated in Phase 1 arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants | 13 [1 to 53]

20. Secondary Outcome: Phase 1: Percentage of Participants Who Were Antitherapeutic Antibody (ATA) Positive, Persistently Positive or Transiently Positive, and Neutralizing Antitherapeutic Antibody (nATA) Positive
Description: ATA positive was defined as participants who have a positive ATA in any postbaseline sample. Transiently ATA positive was defined as participants who have positive ATA in 1 or 2 postbaseline samples. Persistently ATA positive was defined as participants who have positive ATA in more than 2 postbaseline timepoints. Transiently ATA positive was defined as participants who have positive ATA in 1 or 2 postbaseline samples. nATA positive was defined as participants who have at least one positive nATA in any postbaseline ATA positive sample. Here, percentage of participants who were transiently or persistently ATA positive are considered as ATA positive. This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Up to 7 months
Population: Immunogenicity population included participants who received at least 1 dose of study drug and had the baseline immunogenicity sample and at least 1 postbaseline immunogenicity sample assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 +AVD
Number analyzed (Participants) | 8
percentage of participants
  Transiently ATA Positive | 13
  Persistently ATA Positive | 0
  nATA Positive | 0

21. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS per IRF:time from first dose until disease progression per IRF/death due to any cause,whichever occurred first.Participants with no objective progressive disease (PD),did not die,were still on study follow-up at time of analysis were removed from study prior to documentation of PD,PFS was censored on date of last adequate disease assessment before initiation of any non-protocol,alternative therapy.Participants who were on antitumor treatment,other than SCT/radiotherapy,censoring was at last adequate disease assessment before initiation of such alternative treatment.If participant experienced disease progression per IRF/died after initiation of antitumor treatment,other than SCT/radiotherapy,such participant was censored and not considered having PFS.Outcome measure was planned to be assessed for all participant treated at recommended dose in Phase 2.As per SAP,Phase 2 data was summarized and reported in two arms:Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: The safety/efficacy population included participants who received at least 1 dose of any drug in the A+AVD regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
months | NA [NA to NA] — Median and 95% confidence interval (CI) was not estimable due to low number of participants with events. | NA [NA to NA] — Median and 95% confidence interval (CI) was not estimable due to low number of participants with events.

22. Secondary Outcome: Phase 2: Event-free Survival (EFS)
Description: EFS:Time from first dose until any treatment failure:PD per IRF including progression events during follow-up period,failing to complete 6 cycles of treatment due to any reason or death due to any cause,whichever occurred first.EFS per IRF were censored on last adequate disease assessment date per IRF if none of above events occur during study.Participants with antitumor treatment,other than SCT/radiotherapy as part of frontline treatment were censored at last adequate disease assessment before initiation of such alternative treatment.If a participant experienced disease progression per IRF/died after initiation of antitumor treatment,other than SCT/radiotherapy,such participant was censored,and not be considered having EFS.This outcome measure was planned to be assessed for all patients treated at recommended dose in Phase 2.As prespecified in SAP,data for Phase 2 was summarized and reported in two arms:Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: The safety/efficacy population included participants who received at least 1 dose of any drug in the A+AVD regimen. For participants who do not have an objective PD and did not die at the last follow-up, EFS has been censored on the date of last adequate disease assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
months | NA [NA to NA] — Median and 95% CI was not estimable as most of the participants were censored. | NA [NA to NA] — Median and 95% CI was not estimable as most of the participants were censored.

23. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival was defined as time from first dose until death. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive, including study closure. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: The safety/efficacy population included participants who received at least 1 dose of any drug in the A+AVD regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
months | NA [NA to NA] — Median and 95% Cl was not estimable due to low number of participants with events. | NA [NA to NA] — Median and 95% Cl was not estimable due to low number of participants with events.

24. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR per IRF in participants with a response (CR or PR per IRF) was defined as the time from start of the first objective tumor response (CR or PR per IRF) to the first subsequent PD or death due to any cause, whichever occurred first. For patients who did not have an objective PD, did not die and are either still on a study follow-up at the time of the analysis, or were removed from the study prior to documentation of PD, DOR has been censored on the date of last adequate disease assessment. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: Response Evaluable Population=Participants who received at least one dose of study drug, have measurable disease at baseline, and have at least one post-baseline disease assessment (assessments based on investigator assessments or assessments based on an independent review facility). For participants who do not have an objective PD and did not die at the last follow-up, DOR has been censored on the date of last adequate disease assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
months | NA [NA to NA] — Median and 95% confidence interval was not estimable as most of the participants were censored. | NA [NA to NA] — Median and 95% confidence interval was not estimable as most of the participants were censored.

25. Secondary Outcome: Phase 2: Percentage of Participants Receiving Irradiation for HL Following Study Treatment
Description: This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: The safety/efficacy population included participants who received at least 1 dose of any drug in the A+AVD regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 25 [14 to 40] | 24 [14 to 37]

26. Secondary Outcome: Phase 2: Percentage of Participants Who Experienced AEs From the First Dose of Protocol Therapy Through 30 Days After Administration of the Last Dose of Protocol Therapy
Description: as for outcome 25
Time Frame: as for outcome 2
Population: The safety population included participants who had received at least 1 dose of any study drug (A+AVD regimen).
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 100 | 100

27. Secondary Outcome: Phase 2: Percentage of Participants Who Experienced SAEs From the First Dose of Protocol Therapy Through 30 Days After Administration of the Last Dose of Protocol Therapy
Description: as for outcome 25
Time Frame: as for outcome 2
Population: The safety population included participants who had received at least 1 dose of any study drug (A+AVD regimen).
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 45 | 41

28. Secondary Outcome: Phase 2: Percentage of Participants Who Were ATA Positive, Persistently Positive, or Transiently Positive, and nATA Positive
Description: ATA positive was defined as participants who have a positive ATA in any postbaseline sample. Transiently ATA positive was defined as participants who have positive ATA in 1 or 2 postbaseline samples. Persistently ATA positive was defined as participants who have positive ATA in more than 2 postbaseline timepoints. Transiently ATA positive was defined as participants who have positive ATA in 1 or 2 postbaseline samples. nATA positive was defined as participants who have at least one positive nATA in any postbaseline ATA positive sample. Here, percentage of participants who were transiently or persistently ATA positive are considered as ATA positive. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: From first dose until 30 days after the last dose of study drug (up to 7 months)
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants
  Transiently ATA Positive | 6 | 7
  Persistently ATA Positive | 0 | 0
  nATA Positive | 4 | 3

29. Secondary Outcome: Phase 2: Mean Serum Cmax of Brentuximab Vedotin and TAb
Description: as for outcome 25
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 50 | 57
µg/mL
  Cmax of Brentuximab Vedotin at Cycle 1 Day 1 | 23.1 (5.54) | 23.0 (5.21)
  Cmax of Brentuximab Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 34 | 40
  Cmax of Brentuximab Vedotin at Cycle 1 Day 15 | 25.3 (5.12) | 24.9 (4.97)
  Cmax of Brentuximab Vedotin at Cycle 3 Day 1: number analyzed (Participants) | 47 | 55
  Cmax of Brentuximab Vedotin at Cycle 3 Day 1 | 27.4 (6.14) | 27.3 (5.82)
  Cmax of Brentuximab Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 25 | 32
  Cmax of Brentuximab Vedotin at Cycle 3 Day 15 | 25.4 (4.03) | 25.8 (4.81)
  Cmax of TAb Vedotin at Cycle 1 Day 1: number analyzed (Participants) | 48 | 55
  Cmax of TAb Vedotin at Cycle 1 Day 1 | 22.1 (5.34) | 22.4 (5.23)
  Cmax of TAb Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 34 | 40
  Cmax of TAb Vedotin at Cycle 1 Day 15 | 26.5 (9.02) | 26.4 (8.52)
  Cmax of TAb Vedotin at Cycle 3 Day 1: number analyzed (Participants) | 46 | 52
  Cmax of TAb Vedotin at Cycle 3 Day 1 | 29.5 (8.89) | 29.5 (8.44)
  Cmax of TAb Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 25 | 31
  Cmax of TAb Vedotin at Cycle 3 Day 15 | 32.2 (11.0) | 31.4 (10.4)

30. Secondary Outcome: Phase 2: Mean Plasma Cmax of MMAE
Description: as for outcome 25
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 46 | 54
ng/mL
  Cycle 1 Day 1 | 5.49 (2.62) | 5.49 (2.80)
  Cycle 1 Day 15: number analyzed (Participants) | 31 | 37
  Cycle 1 Day 15 | 2.95 (1.66) | 2.81 (1.57)
  Cycle 3 Day 1: number analyzed (Participants) | 45 | 53
  Cycle 3 Day 1 | 1.75 (0.643) | 1.69 (0.635)
  Cycle 3 Day 15: number analyzed (Participants) | 24 | 31
  Cycle 3 Day 15 | 1.74 (0.599) | 1.61 (0.597)

31. Secondary Outcome: Phase 2: Mean Serum AUC0-15d of Brentuximab Vedotin and TAb
Description: as for outcome 25
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 50 | 57
day*µg/mL
  AUC0-15d of Brentuximab Vedotin at Cycle 1 Day 1 | 49.7 (17.2) | 48.8 (16.3)
  AUC0-15d of Brentuximab Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 34 | 40
  AUC0-15d of Brentuximab Vedotin at Cycle 1 Day 15 | 54.9 (22.2) | 54.0 (20.6)
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 1: number analyzed (Participants) | 47 | 54
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 1 | 62.6 (16.9) | 63.9 (18.6)
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 24 | 30
  AUC0-15d of Brentuximab Vedotin at Cycle 3 Day 15 | 60.6 (11.1) | 61.4 (11.5)
  AUC0-15d of TAb at Cycle 1 Day 1: number analyzed (Participants) | 48 | 55
  AUC0-15d of TAb at Cycle 1 Day 1 | 77.2 (18.6) | 77.6 (18.0)
  AUC0-15d of TAb at Cycle 1 Day 15: number analyzed (Participants) | 33 | 39
  AUC0-15d of TAb at Cycle 1 Day 15 | 97.3 (28.7) | 98.1 (27.0)
  AUC0-15d of TAb at Cycle 3 Day 1: number analyzed (Participants) | 46 | 52
  AUC0-15d of TAb at Cycle 3 Day 1 | 119 (30.6) | 120 (29.1)
  AUC0-15d of TAb at Cycle 3 Day 15: number analyzed (Participants) | 23 | 29
  AUC0-15d of TAb at Cycle 3 Day 15 | 124 (21.6) | 125 (24.1)

32. Secondary Outcome: Phase 2: Mean Plasma AUC0-15 of MMAE
Description: as for outcome 25
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 41 | 48
day*ng/mL
  Cycle 1 Day 1 | 31.2 (16.2) | 31.0 (16.8)
  Cycle 1 Day 15: number analyzed (Participants) | 28 | 31
  Cycle 1 Day 15 | 18.4 (11.9) | 17.9 (11.4)
  Cycle 3 Day 1 | 11.5 (5.16) | 11.1 (4.93)
  Cycle 3 Day 15: number analyzed (Participants) | 16 | 20
  Cycle 3 Day 15 | 12.3 (6.12) | 11.3 (5.90)

33. Secondary Outcome: Phase 2: Median Tmax of Brentuximab Vedotin and TAb in Serum
Description: as for outcome 25
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 50 | 57
hour
  Tmax of Brentuximab Vedotin at Cycle 1 Day 1 | 1.03 [0.530 to 164] | 1.00 [0.530 to 164]
  Tmax of Brentuximab Vedotin at Cycle 1 Day 15: number analyzed (Participants) | 34 | 40
  Tmax of Brentuximab Vedotin at Cycle 1 Day 15 | 1.00 [0.500 to 22.7] | 1.00 [0.500 to 22.7]
  Tmax of Brentuximab Vedotin at Cycle 3 Day 1: number analyzed (Participants) | 47 | 55
  Tmax of Brentuximab Vedotin at Cycle 3 Day 1 | 1.00 [0.00 to 23.0] | 1.00 [0.00 to 23.0]
  Tmax of Brentuximab Vedotin at Cycle 3 Day 15: number analyzed (Participants) | 25 | 32
  Tmax of Brentuximab Vedotin at Cycle 3 Day 15 | 1.00 [0.520 to 1.50] | 1.00 [0.520 to 1.50]
  Tmax of TAb at Cycle 1 Day 1: number analyzed (Participants) | 48 | 55
  Tmax of TAb at Cycle 1 Day 1 | 1.01 [0.530 to 20.8] | 1.00 [0.530 to 20.8]
  Tmax of TAb at Cycle 1 Day 15: number analyzed (Participants) | 34 | 40
  Tmax of TAb at Cycle 1 Day 15 | 1.00 [0.500 to 334] | 1.00 [0.500 to 334]
  Tmax of TAb at Cycle 3 Day 1: number analyzed (Participants) | 46 | 52
  Tmax of TAb at Cycle 3 Day 1 | 1.00 [0.00 to 23.3] | 1.00 [0.00 to 23.3]
  Tmax of TAb at Cycle 3 Day 15: number analyzed (Participants) | 25 | 31
  Tmax of TAb at Cycle 3 Day 15 | 1.00 [0.520 to 1.50] | 1.00 [0.520 to 1.50]

34. Secondary Outcome: Phase 2: Median Tmax of MMAE in Plasma
Description: as for outcome 25
Time Frame: Days 1 and 15 of Cycles 1 and 3 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 46 | 54
hour
  Cycle 1 Day 1 | 44.1 [19.7 to 72.0] | 44.4 [19.7 to 72.0]
  Cycle 1 Day 15: number analyzed (Participants) | 31 | 37
  Cycle 1 Day 15 | 42.9 [20.0 to 72.0] | 42.9 [20.0 to 72.0]
  Cycle 3 Day 1: number analyzed (Participants) | 45 | 53
  Cycle 3 Day 1 | 44.9 [20.3 to 71.7] | 45.3 [20.3 to 71.7]
  Cycle 3 Day 15: number analyzed (Participants) | 24 | 31
  Cycle 3 Day 15 | 45.4 [20.0 to 71.7] | 46.0 [20.0 to 71.7]

35. Secondary Outcome: Phase 2: Percentage of Participants Who Experienced Peripheral Neuropathy, Regardless of Seriousness, From the First Dose of Protocol Therapy
Description: Peripheral Neuropathy (PN) was defined by the peripheral neuropathy standardized MedDRA query (SMQ) broad search. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: The safety population included participants who received at least 1 dose of any drug in the A+AVD regimen.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants | 20 | 19

36. Secondary Outcome: Phase 2: Time to Onset and Resolution for All Peripheral Neuropathy Events
Description: Time to onset of first event was defined as time from first dose of study drug to onset of first treatment-emergent PN event. Time to resolution was calculated as the time from onset date to the date of resolution PN (SMQ) event. Participants with multiple resolved events were counted once at the longest time to resolution. Resolution was defined as an event outcome of resolved or resolved with sequelae. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: The safety population included participants who received at least 1 dose of any drug in the A+AVD regimen. Overall number analyzed signifies participants who had peripheral neuropathy were analyzed for this outcome measure, number analyzed are participants with evaluable for the specific category.
Measure: Median (Full Range); unit: weeks
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 12 | 14
weeks
  Time to Onset | 5.93 [0.9 to 19.9] | 5.93 [0.9 to 19.9]
  Time to Resolution: number analyzed (Participants) | 11 | 13
  Time to Resolution | 1.57 [0.3 to 100.3] | 1.57 [0.3 to 100.3]

37. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline Immunoglobulin G Levels at End of Treatment (EOT)
Description: as for outcome 25
Time Frame: Baseline and End of Treatment (Month 7)
Population: Immune Reconstitution Population included participants who received at least 1 dose of study drug and had a sufficient immune reconstitution blood sampling to allow for immune reconstitution evaluation. Number analyzed= number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
g/L
  Baseline: number analyzed (Participants) | 50 | 58
  Baseline | 16.518 (5.5306) | 16.217 (5.2175)
  Change from Baseline at EOT: number analyzed (Participants) | 50 | 57
  Change from Baseline at EOT | -4.822 (4.8964) | -4.675 (4.7204)

38. Secondary Outcome: Phase 1: Percentage of Participants With Low and High ATA Titer Values
Description: High ATA titer was defined as participants who have at least one postbaseline ATA titer less than (>) 25. Low ATA titer was defined as participants whose postbaseline ATA titer are all less than or equal to (<=) 25. This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Up to 6 months
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 8
percentage of participants
  ATA Titer low | 13
  ATA Titer High | 0

39. Secondary Outcome: Phase 2: Percentage of Participants With Low and High ATA Titer Values
Description: High ATA titer was defined as participants who have at least one postbaseline ATA titer >25. Low ATA titer was defined as participants whose postbaseline ATA titer are all <=25. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 6 months
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants
  ATA Titer Low | 6 | 7
  ATA Titer High | 0 | 0

40. Secondary Outcome: Phase 1: Mean Cmax of Brentuximab Vedotin in ATA Positive and ATA Negative Participants
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Cycle 1 and 3: Days 1 and 15 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 8
µg/mL
  ATA Positive: Cycle 1 Day 1: number analyzed (Participants) | 1
  ATA Positive: Cycle 1 Day 1 | 23.3 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Positive: Cycle 1 Day 15: number analyzed (Participants) | 1
  ATA Positive: Cycle 1 Day 15 | 21.1 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Positive: Cycle 3 Day 1: number analyzed (Participants) | 1
  ATA Positive: Cycle 3 Day 1 | 23.1 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Positive: Cycle 3 Day 15: number analyzed (Participants) | 1
  ATA Positive: Cycle 3 Day 15 | 21.6 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Negative: Cycle 1 Day 1: number analyzed (Participants) | 6
  ATA Negative: Cycle 1 Day 1 | 22.5 (1.62)
  ATA Negative: Cycle 1 Day 15: number analyzed (Participants) | 5
  ATA Negative: Cycle 1 Day 15 | 23.5 (4.17)
  ATA Negative: Cycle 3 Day 1: number analyzed (Participants) | 7
  ATA Negative: Cycle 3 Day 1 | 27.2 (3.62)
  ATA Negative: Cycle 3 Day 15: number analyzed (Participants) | 6
  ATA Negative: Cycle 3 Day 15 | 28.3 (7.32)

41. Secondary Outcome: Phase 1: Mean AUC 0-15d of Brentuximab Vedotin in ATA Positive and ATA Negative Participants
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Cycle 1 and 3: Days 1 and 15 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 8
day*µg/mL
  ATA Positive: Cycle 1 Day 1: number analyzed (Participants) | 1
  ATA Positive: Cycle 1 Day 1 | 42.4 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Positive: Cycle 1 Day 15: number analyzed (Participants) | 1
  ATA Positive: Cycle 1 Day 15 | 50.0 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Positive: Cycle 3 Day 1: number analyzed (Participants) | 1
  ATA Positive: Cycle 3 Day 1 | 56.6 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Positive: Cycle 3 Day 15: number analyzed (Participants) | 1
  ATA Positive: Cycle 3 Day 15 | 63.0 (NA) — The standard deviation was not estimable for one participant with event.
  ATA Negative: Cycle 1 Day 1: number analyzed (Participants) | 6
  ATA Negative: Cycle 1 Day 1 | 42.2 (3.40)
  ATA Negative: Cycle 1 Day 15: number analyzed (Participants) | 5
  ATA Negative: Cycle 1 Day 15 | 48.6 (6.48)
  ATA Negative: Cycle 3 Day 1: number analyzed (Participants) | 6
  ATA Negative: Cycle 3 Day 1 | 75.4 (29.46)
  ATA Negative: Cycle 3 Day 15: number analyzed (Participants) | 5
  ATA Negative: Cycle 3 Day 15 | 65.1 (15.06)

42. Secondary Outcome: Phase 1: Percentage of Participants Achieving CR Per IRF Assessment Per IWG Criteria in ATA Positive and ATA Negative Participants
Description: CR was defined as the disappearance of all evidence of disease as assessed by IRF as per IWG Criteria. The data is reported per ATA status as categories. This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Up to 24 months
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 8
percentage of participants
  ATA Negative who Achieved CR: number analyzed (Participants) | 7
  ATA Negative who Achieved CR | 86 [42 to 100]
  Transiently ATA Positive who Achieved CR: number analyzed (Participants) | 1
  Transiently ATA Positive who Achieved CR | 100 [3 to 100]

43. Secondary Outcome: Phase 1: Number of ATA Positive and ATA Negative Participants With AEs and SAEs
Description: This outcome measure is planned to be assessed only for participants treated in Phase 1 arm.
Time Frame: Up to 24 months
Population: The Safety Population included participants who received at least 1 dose of any drug in the A+AVD regimen, with data available for analyses. Data is reported as per ATA positive and negative status.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD: Brentuximab vedotin 48 mg/m^2 (A), intravenous infusion, once on Days 1 and 15 of each 28-day cycle approximately 1 hour after administration of doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (AVD), intravenous infusion, once on Days 1 and 15 of each 28-day cycle for up to 6 cycles. Participants who received at least one dose of study in Phase 1 and continued to receive the study drug in Phase 2 were included in this arm group.
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 8
Participants
  ATA Negative: AEs: number analyzed (Participants) | 7
  ATA Negative: AEs | 7
  ATA Positive: AEs: number analyzed (Participants) | 1
  ATA Positive: AEs | 1
  ATA Negative: SAEs: number analyzed (Participants) | 7
  ATA Negative: SAEs | 0
  ATA Positive: SAEs: number analyzed (Participants) | 1
  ATA Positive: SAEs | 1

44. Secondary Outcome: Phase 2: Mean Cmax of Brentuximab Vedotin in ATA Positive and ATA Negative Participants
Description: as for outcome 25
Time Frame: Cycle 1-3: Days 1 and 15 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
µg/mL
  ATA Positive: Cycle 1 Day 1: number analyzed (Participants) | 3 | 4
  ATA Positive: Cycle 1 Day 1 | 27.8 (8.56) | 26.7 (7.34)
  ATA Positive: Cycle 1 Day 15: number analyzed (Participants) | 3 | 4
  ATA Positive: Cycle 1 Day 15 | 23.3 (6.88) | 22.7 (5.72)
  ATA Positive: Cycle 3 Day 1: number analyzed (Participants) | 2 | 3
  ATA Positive: Cycle 3 Day 1 | 22.0 (2.92) | 22.4 (2.15)
  ATA Positive: Cycle 3 Day 15: number analyzed (Participants) | 2 | 3
  ATA Positive: Cycle 3 Day 15 | 25.6 (7.93) | 24.2 (6.07)
  ATA Negative: Cycle 1 Day 1: number analyzed (Participants) | 47 | 53
  ATA Negative: Cycle 1 Day 1 | 22.8 (5.29) | 22.7 (5.00)
  ATA Negative: Cycle 1 Day 15: number analyzed (Participants) | 31 | 36
  ATA Negative: Cycle 1 Day 15 | 25.4 (5.02) | 25.2 (4.91)
  ATA Negative: Cycle 3 Day 1: number analyzed (Participants) | 45 | 52
  ATA Negative: Cycle 3 Day 1 | 27.7 (6.14) | 27.6 (5.84)
  ATA Negative: Cycle 3 Day 15: number analyzed (Participants) | 23 | 29
  ATA Negative: Cycle 3 Day 15 | 25.4 (3.85) | 26.0 (4.76)

45. Secondary Outcome: Phase 2: Mean AUC 0-15 of Brentuximab Vedotin in ATA Positive and ATA Negative Participants
Description: as for outcome 25
Time Frame: Cycle 1-3: Days 1 and 15 pre-infusion and up to 30 minutes after the end of infusion (Cycle length=28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
day*µg/mL
  ATA Positive: Cycle 1 Day 1: number analyzed (Participants) | 3 | 4
  ATA Positive: Cycle 1 Day 1 | 51.6 (17.17) | 49.3 (14.75)
  ATA Positive: Cycle 1 Day 15: number analyzed (Participants) | 3 | 4
  ATA Positive: Cycle 1 Day 15 | 45.6 (38.87) | 46.7 (31.81)
  ATA Positive: Cycle 3 Day 1: number analyzed (Participants) | 2 | 3
  ATA Positive: Cycle 3 Day 1 | 53.7 (10.16) | 54.6 (7.38)
  ATA Positive: Cycle 3 Day 15: number analyzed (Participants) | 2 | 3
  ATA Positive: Cycle 3 Day 15 | 57.2 (12.37) | 59.1 (9.38)
  ATA Negative: Cycle 1 Day 1: number analyzed (Participants) | 47 | 53
  ATA Negative: Cycle 1 Day 1 | 49.6 (17.41) | 48.8 (16.58)
  ATA Negative: Cycle 1 Day 15: number analyzed (Participants) | 31 | 36
  ATA Negative: Cycle 1 Day 15 | 55.8 (20.77) | 54.8 (19.52)
  ATA Negative: Cycle 3 Day 1: number analyzed (Participants) | 45 | 51
  ATA Negative: Cycle 3 Day 1 | 63.0 (17.10) | 64.4 (18.99)
  ATA Negative: Cycle 3 Day 15: number analyzed (Participants) | 22 | 27
  ATA Negative: Cycle 3 Day 15 | 60.9 (11.23) | 61.7 (11.81)

46. Secondary Outcome: Phase 2: Percentage of Participants Achieving CR Per IRF Assessment Per IWG Criteria in ATA Positive and ATA Negative Participants
Description: CR is defined as the disappearance of all evidence of disease as assessed by IRF as per IWG Criteria. This outcome measure was planned to be assessed only for all participants treated at the recommended dose in Phase 2. As prespecified in SAP, data for Phase 2 was summarized and reported in two arms: Phase 2 and Phase 1 + Phase 2.
Time Frame: Up to 24 months
Population: Immunogenicity Population included participants who received at least 1 dose of study drug and had the baseline immunogenicity sample and at least 1 postbaseline immunogenicity sample assessment. Number analyzed is the number of participants analyzed for the specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
percentage of participants
  ATA Negative: number analyzed (Participants) | 48 | 55
  ATA Negative | 75 [60 to 86] | 76 [63 to 87]
  Transiently ATA Positive: number analyzed (Participants) | 3 | 4
  Transiently ATA Positive | 67 [9 to 99] | 75 [19 to 99]

47. Secondary Outcome: Phase 2: Number of ATA Positive and ATA Negative Participants With AEs and SAEs
Description: as for outcome 25
Time Frame: Up to 24 months
Population: The Safety Population included participants who received at least 1 dose of any drug in the A+AVD regimen. Data is reported as per ATA positive and negative status.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 51 | 59
Participants
  ATA Negative: AEs: number analyzed (Participants) | 48 | 55
  ATA Negative: AEs | 48 | 55
  ATA Positive: AEs: number analyzed (Participants) | 3 | 4
  ATA Positive: AEs | 3 | 4
  ATA Negative: SAEs: number analyzed (Participants) | 48 | 55
  ATA Negative: SAEs | 21 | 21
  ATA Positive: SAEs: number analyzed (Participants) | 3 | 4
  ATA Positive: SAEs | 2 | 3

48. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in Immunoglobulin M at the End of Treatment (EOT)
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: Immune Reconstitution Population included participants who received at least 1 dose of study drug and had a sufficient immune reconstitution blood sampling to allow for immune reconstitution evaluation, with data available for analyses. Number analyzed is number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 48 | 56
g/L
  Baseline | 1.275 (0.5065) | 1.261 (0.4824)
  Change at EOT (Month 7): number analyzed (Participants) | 46 | 53
  Change at EOT (Month 7) | -0.345 (0.5942) | -0.375 (0.5766)

49. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in Immunoglobulin A at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: Immune Reconstitution Population included participants who received at least 1 dose of study drug and had a sufficient immune reconstitution blood sampling to allow for immune reconstitution evaluation. Overall number analyzed are the participants with data available for analyses. Number analyzed= number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 49 | 57
g/L
  Baseline | 2.708 (1.2379) | 2.671 (1.1879)
  Change from Baseline at EOT: number analyzed (Participants) | 47 | 54
  Change from Baseline at EOT | -0.195 (1.0479) | -0.125 (1.0844)

50. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in Tetanus at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: Immune Reconstitution Population included participants who received at least 1 dose of study drug and had a sufficient immune reconstitution blood sampling to allow for immune reconstitution evaluation. Overall number analyzed are the number of participants with data available for analyses. Number analyzed =number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: (IU)/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 48 | 56
(IU)/mL
  Baseline | 1.636 (2.5600) | 1.935 (3.0358)
  Change from Baseline at EOT: number analyzed (Participants) | 42 | 49
  Change from Baseline at EOT | -0.648 (1.3412) | -0.914 (2.2679)

51. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in Haemophilus Influenzae B Antibody, IgG at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: Immune Reconstitution Population included participants who received at least 1 dose of study drug and had a sufficient immune reconstitution blood sampling to allow for immune reconstitution evaluation. Overall number analyzed are the number of participants with data available for analyses. Number analyzed= number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 50 | 58
µg/mL
  Baseline | 10.39 (27.017) | 9.50 (25.167)
  Change from Baseline at EOT: number analyzed (Participants) | 49 | 55
  Change from Baseline at EOT | -7.00 (24.258) | -6.03 (23.160)

52. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline Poliovirus Antibodies Ratio at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 50 | 58
ratio
  Baseline: Type I | 0.02447 (0.027568) | 0.02373 (0.028092)
  EOT: Type I: number analyzed (Participants) | 50 | 56
  EOT: Type I | 0.00913 (0.024223) | 0.00845 (0.023091)
  Baseline: Type III | 0.03641 (0.036709) | 0.03432 (0.036653)
  EOT: Type III: number analyzed (Participants) | 50 | 56
  EOT: Type III | 0.01141 (0.029889) | 0.01013 (0.028461)

53. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline Total Immunoglobulin at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 48 | 56
mg/dl
  Baseline | 2086.6 (615.62) | 2045.1 (583.04)
  Change from Baseline at EOT: number analyzed (Participants) | 46 | 56
  Change from Baseline at EOT | -582.3 (565.52) | -556.3 (553.97)

54. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in Peripheral Blood CD34+A at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 38 | 44
µL
  Baseline | 4.182 (4.1227) | 3.917 (3.8917)
  Change from Baseline at EOT: number analyzed (Participants) | 29 | 34
  Change from Baseline at EOT | -1.512 (4.7075) | -1.456 (4.3472)

55. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in Total Lymphocyte Count at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: Immune Reconstitution Population included participants who received at least 1 dose of study drug and had a sufficient immune reconstitution blood sampling to allow for immune reconstitution evaluation.
Measure: Mean (Standard Deviation); unit: 10^9 lymphocytes/L
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 49 | 57
10^9 lymphocytes/L
  Baseline | 1.8022 (0.95206) | 1.7408 (0.91394)
  Change from Baseline at EOT: number analyzed (Participants) | 48 | 56
  Change from Baseline at EOT | 0.6736 (3.77611) | 0.5965 (3.50121)

56. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in the Percentage of CD4+ (CD4+CD45RA-CD197- and CD4+CD45RA+CD197+) Subset of Cells at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: percentage of CD4+ subset cells
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 32 | 39
percentage of CD4+ subset cells
  Baseline: CD4+CD45RA-CD197- | 28.0 (12.76) | 29.0 (13.42)
  Change from Baseline at EOT: CD4+CD45RA-CD197-: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD4+CD45RA-CD197- | -5.0 (17.72) | -5.1 (16.44)
  Baseline: CD4+CD45RA-CD197+ | 23.7 (14.33) | 22.3 (13.86)
  Change from Baseline at EOT: CD4+CD45RA-CD197+: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD4+CD45RA-CD197+ | 13.0 (14.14) | 12.6 (13.21)
  Baseline: CD4+CD45RA+CD197- | 2.9 (3.41) | 3.1 (3.22)
  Change from Baseline at EOT: CD4+CD45RA+CD197-: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD4+CD45RA+CD197- | -0.7 (2.25) | -0.7 (2.41)
  Baseline: CD4+CD45RA+CD197+ | 46.2 (14.44) | 46.3 (14.89)
  Change from Baseline at EOT: CD4+CD45RA+CD197+: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD4+CD45RA+CD197+ | -7.2 (11.60) | -6.8 (11.04)

57. Secondary Outcome: Phase 2: Immune Reconstitution-Change From Baseline in the Percentage of CD8+ (CD8+CD45RA-CD197- and CD8+CD45RA-CD197+) Subset of Cells at EOT
Description: as for outcome 25
Time Frame: Baseline, EOT [Month 7]
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: percentage of CD8+ subset cells
Arm/Group | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 1 + Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
Number analyzed (Participants) | 32 | 39
percentage of CD8+ subset cells
  Baseline: CD8+CD45RA-CD197- | 39.9 (19.32) | 40.6 (20.00)
  Change from Baseline at EOT: CD8+CD45RA-CD197-: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD8+CD45RA-CD197- | -11.5 (13.85) | -11.0 (14.33)
  Baseline: CD8+CD45RA-CD197+: number analyzed (Participants) | 28 | 35
  Baseline: CD8+CD45RA-CD197+ | 2.4 (1.81) | 2.3 (1.76)
  Change from Baseline at EOT: CD8+CD45RA-CD197+: number analyzed (Participants) | 20 | 26
  Change from Baseline at EOT: CD8+CD45RA-CD197+ | 1.6 (2.52) | 2.1 (3.08)
  Baseline: CD8+CD45RA+CD197- | 25.9 (15.43) | 25.8 (14.60)
  Change from Baseline at EOT: CD8+CD45RA+CD197-: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD8+CD45RA+CD197- | -6.0 (11.27) | -6.5 (11.83)
  Baseline: CD8+CD45RA+CD197+ | 31.3 (18.00) | 30.8 (18.53)
  Change from Baseline at EOT: CD8+CD45RA+CD197+: number analyzed (Participants) | 23 | 29
  Change from Baseline at EOT: CD8+CD45RA+CD197+ | 15.7 (11.48) | 15.4 (12.15)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to data cut -off date: 24 September 2021 (Up to approximately 4 years)
Description: The Safety Population included participants who received at least 1 dose of any drug in the A+AVD regimen. Data is reported in 2 arms: Phase 1 includes participants who received at least one dose of study drug in Phase 1 and continued to Phase 2 to receive the same drug; Phase 2 included participants who were enrolled directly in Phase 2 to receive the study drug at recommended dose in Phase 2 only.
Arm/Group | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/8 | 23/51
Other Adverse Events (participants affected / at risk) | 8/8 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD (N=8) | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 9
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Brentuximab Vedotin 48 mg/m^2 + AVD (N=8) | Phase 2: Brentuximab Vedotin 48 mg/m^2 + AVD (N=51)
Vomiting (Gastrointestinal disorders) | 8 | 42
Nausea (Gastrointestinal disorders) | 8 | 36
Abdominal pain (Gastrointestinal disorders) | 2 | 21
Stomatitis (Gastrointestinal disorders) | 4 | 21
Constipation (Gastrointestinal disorders) | 4 | 17
Diarrhoea (Gastrointestinal disorders) | 4 | 10
Abdominal pain upper (Gastrointestinal disorders) | 8 | 7
Oral pain (Gastrointestinal disorders) | 1 | 7
Odynophagia (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 20
Fatigue (General disorders) | 3 | 9
Asthenia (General disorders) | 5 | 3
Pain (General disorders) | 0 | 6
Catheter site pain (General disorders) | 1 | 3
Chills (General disorders) | 1 | 2
Influenza like illness (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 20
Anaemia (Blood and lymphatic system disorders) | 1 | 12
Leukopenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
White blood cell count decreased (Investigations) | 5 | 20
Neutrophil count decreased (Investigations) | 4 | 18
Weight decreased (Investigations) | 1 | 12
Lymphocyte count decreased (Investigations) | 0 | 7
Polymerase chain reaction positive (Investigations) | 1 | 3
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Rhinitis (Infections and infestations) | 3 | 7
Conjunctivitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 5
Oral herpes (Infections and infestations) | 1 | 4
Pharyngitis (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 5 | 14
Dizziness (Nervous system disorders) | 1 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 12
Dehydration (Metabolism and nutrition disorders) | 0 | 5
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 5
Palpitations (Cardiac disorders) | 1 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 6
Insomnia (Psychiatric disorders) | 1 | 3
Hyperaemia (Vascular disorders) | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT02979522/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT02979522/SAP_001.pdf